CLINICAL TRIAL: NCT05179382
Title: Integrated Analysis of Autonomic, Cardiovascular and Respiratory Parameters in Recovery After Physical Exercise With and Without Water Ingestion: Crossover Non-randomized Clinical Test
Brief Title: Integrated Analysis in Recovery After Exercise With and Without Hydration.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luiz Carlos Marques Vanderlei (Other)
Responsible Party: Sponsor-Investigator, Luiz Carlos Marques Vanderlei, PhD, Universidade Estadual Paulista Júlio de Mesquita Filho
Organization: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 38152620500005402
Record Dates: First submitted 2021-12-17; First posted 2022-01-05 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control protocol (Active Comparator): The control protocol will consist of an initial 10 minutes of rest, followed by 90 minutes of aerobic activity and 60 minutes of the final recovery. Hydration will not be allowed throughout the protocol.
  Interventions: Other: Control protocol
- Hydration protocol (Experimental): This intervention will consist of an initial 10 minutes of rest, followed by 90 minutes of aerobic activity and 60 minutes of the final recovery. In this protocol, volunteers will be hydrated with mineral water from the 15th minute of exercise until the end of recovery.
  Interventions: Other: Hydration protocol

INTERVENTIONS:
Other: Control protocol — I.10 minutes of initial rest in the supine position; II. 90 minutes of treadmill aerobic exercise at an intensity of 60% of the vo2 peak; IV. 60 minutes of passive recovery in the supine position.
  Arms: Control protocol
Other: Hydration protocol — I.10 minutes of initial rest in the supine position; II. 90 minutes of treadmill aerobic exercise at an intensity of 60% of the vo2 peak; IV. 60 minutes of passive recovery in the supine position. V. Water ingestion distributed in 10 equal portions, administered at regular intervals of 15 minutes from the 15th minute of exercise until the end of the recovery period.
  Arms: Hydration protocol

SUMMARY:
This study aims to evaluate post-exercise recovery in healthy young men submitted to a prolonged exercise protocol of submaximal intensity with or without water intake, from the integrated analysis of autonomic (heart rate variability indices), cardiovascular outcomes (systolic blood pressure, diastolic blood pressure and heart rate) and respiratory (oxygen saturation and respiratory frequency). In addition, it will also be evaluated whether the proposed model is able to estimate the number of individuals undergoing hydration that have better recovery.

ELIGIBILITY:
Inclusion Criteria:

* Include healthy and male individuals, age between 18 and 25 years and physically active.

Exclusion Criteria:

* Volunteers with at least one of the following characteristics will be excluded: smoking, use of drugs that influence the autonomic activity of the heart, alcoholics, people with known metabolic and/or endocrine disorders, and sedentary individuals, insufficiently active and very active.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Acute evaluation during interventions
  Will occur indirectly, using a stethoscope and an aneroid sphygmomanometer in the left arm. The indicated values will be registered in an individual form. To avoid errors in the determination of blood pressures in volunteers, a single evaluator will measure these variables throughout the experimental procedure. Data will be collected at the end of the 10 minutes of initial rest and at minutes 30, 60 and 90 during exercise on the treadmill, as well as will be collected at minutes 1, 3, 5, 7, 10, 20, 30, 40, 50 and 60 of recovery.
Heart Rate | Acute evaluation during interventions
  The heart rate will be captured beat by beat using the Polar RS800CX frequency meter, equipment previously validated to capture this parameter. Data will be collected at the end of the 10 minutes of initial rest and at minutes 30, 60 and 90 during exercise on the treadmill, as well as will be collected at minutes 1, 3, 5, 7, 10, 20, 30, 40, 50 and 60 of recovery.
Respiratory Rate | Acute evaluation during interventions
  The measurements will be performed by counting the breaths for one minute without the volunteer being aware of the process, so that the usual breathing characteristics are not modified. Data will be collected at the end of the 10 minutes of initial rest as well as will be collected at minutes 1, 3, 5, 7, 10, 20, 30, 40, 50 and 60 of recovery.
Peripheral oxygen saturation | Acute evaluation during interventions
  Will be checked using a pulse oximeter. A pulse oximeter is a device that provides blood saturation readings, evaluating the absorption behavior of oxyhemoglobin and deoxyhemoglobin in relation to the lengths of red and infrared light. Data will be collected at the end of the 10 minutes of initial rest and at minutes 30, 60 and 90 during exercise on the treadmill, as well as will be collected at minutes 1, 3, 5, 7, 10, 20, 30, 40, 50 and 60 of recovery.
Autonomic Modulation - rMSSD index | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. The rMSSD index corresponds to the root-mean square of differences between adjacent normal RR intervals in a time interval, expressed in milliseconds.
Autonomic Modulation - SDNN index | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. The SDNN index corresponds to the standard deviation of all normal RR intervals recorded in a time interval, expressed in milliseconds.
Autonomic Modulation - LF index | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. The LF index is the low-frequency component of the oscillatory components of heart rate variability, and ranges from 0.04 to 0.15 Hz.
Autonomic Modulation - HF index | Acute evaluation during interventions
  he data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. The HF index is the high-frequency component of the oscillatory components of heart rate variability, and ranges from 0.15 to 0.4 Hz.
Autonomic Modulation - SD1 index | Acute evaluation during interventions
  he data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. The SD1 index corresponds to the dispersion of points perpendicular to the line of identity of the ellipse obtained from the Poincaré plot. Expressed in milliseconds.
Autonomic Modulation - SD2 index | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. The SD2 index corresponds to the dispersion of points along the line of identity of the ellipse obtained from the Poincaré plot. Expressed in milliseconds.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Carlos M Vanderlei, PhD, Study Director — Professor
Locations (1):
- Universidade Estadual Paulista Júlio de Mesquita Filho, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No